CLINICAL TRIAL: NCT02410642
Title: Effects of Cardiopulmonary Bypass on Urinary Secretion of NAG
Brief Title: NAG-excretion During Cardiopulmonary Bypass
Acronym: CPBNAG
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lukas Lannemyr, MD, Sahlgrenska University Hospital
Other Study IDs: SahlgrenskaUHThoraxLL2
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Renal Impairment
Keywords: cardiopulmonary bypass
MeSH Terms: conditions — Renal Insufficiency | interventions — Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cardiopulmonary bypass — Routine use of cardiopulmonary bypass as needed during cardiac surgery

SUMMARY:
NAG is a protein excreted in urine in cases of tubular damage, and is considered a biomarker of kidney injury. Elevated urinary NAG is seen after cardiac surgery, but the clinical significance, pattern of excretion and links to perioperative factors are poorly described. We plan a study of the pattern of NAG-excretion during cardiac surgery with cardiopulmonary bypass, and explore possible associated variables.

DETAILED DESCRIPTION:
The standard biomarker of AKI, serum creatinine, has poor specificity and sensitivity in the early phases of renal injury. Since the therapeutic window is likely to be in the earlier stages before renal injury is manifest, there is a need for novel diagnostic methods. In the recent years, several new biomarkers of kidney injury have been introduced. To date, none has proven outstanding regarding precision in early detection of AKI. NAG (N-acetyl-b-D-glucosaminidase) is a lysosomal enzyme with high molecular weight. Due to its size, NAG does not normally pass the glomerulus apparatus, but urine levels are elevated after tubulus damage. NAG excretion in urine is seen in AKI after cardiac surgery, exposure to nephrotoxic agents and after renal transplantation. However, its role in clinical decision-making is yet to be established.

We aim to study the excretion pattern of urinary NAG during and after cardiac surgery with cardiopulmonary bypass. Association with perioperative variables will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Expected cardiopulmonary bypass time exceeding 60 minutes
* Elective surgery

Exclusion Criteria:

* End-stage kidney disease with dialysis
* Ongoing treatment with nephrotoxic antibiotic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients scheduled for complex cardiac surgery
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Urinary NAG secretion | 24 hours
  Secretion pattern of NAG

SECONDARY OUTCOMES:
Development of AKI (acute kidney injury) according to AKIN criteria | 72 hours
  Development of AKI (acute kidney injury) according to AKIN criteria

OTHER OUTCOMES:
Perioperative factors influencing NAG-secretion | 24 hours
  Multivariate analysis of factors that might influence NAG-excretion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of thoracic anesthesia, Sahlgrenska University Hospital, Gothenburg, Sweden